CLINICAL TRIAL: NCT03603054
Title: Analysing the Immediate Effects of Sciatic Nerve Mobilization on the Range of Cervical Mobility and on the Myofascial Trigger Points of the Cervical Muscles. Pilot Study.
Brief Title: The Effect of Lower Limbs Neural Mobilization in Subjects With Cervical Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Roser Bel-lan Roldan, physiotherapist, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPC.EPP.02.18
Record Dates: First submitted 2018-07-12; First posted 2018-07-27 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-07

CONDITIONS: Neck Pain
Keywords: Neck pain; Neural mobilization; Myofascial trigger point; Sciatic nerve
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: The study sample will be randomly divide into 2 groups, a control group subject to a placebo technique and an intervention group subject to an active mobilization of the sciatic nerve.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active neck mobilization (Active Comparator): The subjects, who were randomly allocated to group active neurodynamic mobilization group, will receive the active sciatic nerve mobilization intervention. The subject will be instructed to do a a modification of the slump. The procedure will be performed 1 minute with each leg, two times, the subjects will rest one minute between each mobilization and between series.
  Interventions: Other: Active neck mobilization
- Active Mobilization of the Sciatic nerve (Experimental): The subjects, who were randomly allocated to group active neurodynamic mobilization group, will receive the active sciatic nerve mobilization intervention. The subject will be instructed to do a a modification of the slump. The procedure will be performed 1 minute with each leg, two times, the subjects will rest one minute between each mobilization and between series.
  Interventions: Other: Active Mobilization of the sciatic nerve

INTERVENTIONS:
Other: Active neck mobilization — The subjects, receive an active neck mobilization intervention.
  Arms: Active neck mobilization
Other: Active Mobilization of the sciatic nerve — The subjects, receive an active sciatic nerve mobilization intervention.
  Arms: Active Mobilization of the Sciatic nerve

SUMMARY:
No studies have investigated the effects of a Sciatic nerve mobilization in subjects with neck pain. This study aims to determine the immediate effects of a lower limbs neural mobilization on cervical range of motion and on the perception of pain in the most common trigger points located in the cervical musculature.

DETAILED DESCRIPTION:
A convenience sample will be used to obtain subjects The subjects will be recruited through posted advertisements on social networks. The inclusion and exclusion criteria will be applied to the volunteers. The sample wil comprise university students and administrative workers with neck pain. The subjects will be screened by a screening questionnaire and all of them, they will be required to sign an inform consent before participating to the study. After signing it, they will be randomly divide into control group subject to a placebo technique and the intervention group subject to an active mobilization of the sciatic nerve.

To assess changes in cervical articular range, will be used, a cervical goniometer (CROM) and for changes in pressure pain threshold of the trigger points will be used a mechanical algometer. Furthermore, to asses changes in pain perception will be used a visual numerical scale. The statistical analysis will be performed using the statistical program SPSS 25.0, comparing the results between both groups.

ELIGIBILITY:
Inclusion Criteria:

* To spend more than 3 hours at the computer.
* To have or have had neck pain during the last 3 weeks.

Exclusion Criteria:

* To have had traumatisms, traffic accidents and surgeries in the last 2 months.
* To have taken any analgesic tablets before the treatment.
* To be in a physiotherapy treatment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Pain level at rest | Change from baseline in Visual Analog Scale at 2 minutes after intervention
  A Visual Analog Scale, will be used for recording level of pain at rest. The VAS evaluates levels of pain intensity using an 10-point scale (range 0-10), with 0 being classified as "no sensation" and 10 "pain as bad as could be".

SECONDARY OUTCOMES:
Cervical Range of Motion (CROM) | Before intervention and 2 minutes after
  The Cervical Range of Motion (CROM) device will be used to measure the cervical range of motion, including flexion, extension, lateral flexion and rotation.
Mechanical pressure Algometer | Before intervention and 2 minutes after
  The Mechanical pressure Algometer will be used to measure changes in pain threshold of sensitive points located in the cervical musculature.
Vernier caliper | Before intervention and 2 minutes after
  The Vernier caliper will be used to measure the active opening of the mouth.
The Neck Disability Index, Spanish version | Before intervention
  The Neck Disability Index questionnaire is a reliable instrument to assess functional disability in neck pain patients. Will be used to assess the subjects' perceived disability level and how their neck pain affect to their daily live.
  Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. All the points can be summed to a total score. The test can be interpretated as a raw score, with a maximum score of 50, or as a percentage.
  0 points or 0% means : no activity limitations , 50 points or 100% means complete activity limitation.
Hours of daily use of display screens | Before intervention
  The subjects will be asked at the beginning of the study about how many hours they spend using display screens daily.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Hernández-Sánchez, PhD-PT, Study Director — Universidad Miguel Hernandez de Elche; Carlos Lozano-Quijada, PhD-PT, Study Director — Universidad Miguel Hernandez de Elche; Roser Bel-lan, PT, Principal Investigator — Universidad Miguel Hernandez de Elche
Locations (1):
- Miguel Hernandez University, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No